CLINICAL TRIAL: NCT00371189
Title: A Phase I Randomized, Controlled, Dosage-Escalation Trial to Evaluate the Immunogenicity, Safety, and Reactogenicity of an Adenovirus Type 35 Based Circumsporozoite Malaria Vaccine in Healthy Adults 18 to 45 Years of Age
Brief Title: Adenovirus Vaccine for Malaria
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 05-0050; N01AI80007C
Record Dates: First submitted 2006-08-31; First posted 2006-09-01 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-06

CONDITIONS: Plasmodium Falciparum Infection
Keywords: circumsporozoite, malaria, vaccine
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- Group C: Ad35.CS.01-10^10 vp/ml (Experimental): 15 subjects will receive dosage 10^10 vp/mL; 3 subjects will receive placebo.
  Interventions: Drug: Placebo; Biological: Ad35.CS.01 Circumsporozoite Malaria Vaccine
- Group D: Ad35.CS.01-10^11 vp/ml (Experimental): 15 subjects will receive dosage 10^11 vp/mL; 3 subjects will receive placebo.
  Interventions: Drug: Placebo; Biological: Ad35.CS.01 Circumsporozoite Malaria Vaccine
- Group A: Ad35.CS.01-10^8 vp/ml (Experimental): 15 subjects will receive dosage 10^8 vp/mL; 3 subjects will receive placebo.
  Interventions: Drug: Placebo; Biological: Ad35.CS.01 Circumsporozoite Malaria Vaccine
- Group B: Ad35.CS.01-10^9 vp/ml (Experimental): 15 subjects will receive dosage 10^9 vp/mL; 3 subjects will receive placebo.
  Interventions: Drug: Placebo; Biological: Ad35.CS.01 Circumsporozoite Malaria Vaccine

INTERVENTIONS:
Drug: Placebo — Normal saline.
Biological: Ad35.CS.01 Circumsporozoite Malaria Vaccine — Adenovirus Type 35 Circumsporozoite Malaria Vaccine (Ad35.CS.01); administered at 0, 1, and 6 months; dosage levels: 10^8 viral particles (vp)/mL, 10^9 vp/mL, 10^10 vp/mL and 10^11 vp/mL.

SUMMARY:
Malaria is caused by a parasite carried by a mosquito. Currently, there is no vaccine licensed to prevent malaria. The purpose of this study is to find the most effective and safest dose of an experimental vaccine for the treatment of malaria. Participants will include 72 healthy adults, ages18 to 45, enrolled at Vanderbilt University Medical Center and Stanford University. Volunteers will receive 3 doses of either the malaria vaccine or placebo (contains no vaccine) by injection into a muscle at 0, 1 and 6 months. Investigators will evaluate how the body responds to increasing dosage strengths of the vaccine. Study procedures include physical exam, multiple blood draws, and completion of a memory aid (diary). Each participant will be actively involved in the study for about 12 months. Then, an annual phone call will be made to check for any serious illness events for a period of 5 years.

DETAILED DESCRIPTION:
Malaria currently represents one of the most prevalent infections in tropical and subtropical areas throughout the world. Each year, malaria affects around 300 million people and kills 1 to 3 million people in developing countries. The widespread occurrence and the growing incidence of malaria are a consequence of the increasing numbers of drug-resistant parasites and insecticide-resistant parasite vectors. Other factors include environmental and climatic changes, civil disturbances and increased mobility of populations. It is hypothesized that the Ad35.CS.01 vaccine will prevent the Plasmodium (P.) falciparum parasite, which causes malaria, from entering and developing within the liver of those who become infected. Ad35.CS.01 would therefore be expected to reduce malaria-attributable morbidity and mortality. The purpose of this phase I, randomized, controlled, dosage-escalation trial is to evaluate the immunogenicity, safety, and reactogenicity of an Adenovirus Type 35 based circumsporozoite malaria vaccine in 72 healthy adults, 18 to 45 years of age, in the United States. Subjects will be randomized in a 5:1 ratio to receive 3 doses of the Adenovirus Type 35 circumsporozoite malaria vaccine (Ad35.CS.01) or normal saline placebo control by the intramuscular route at 0, 1 and 6 months. The safety, reactogenicity, and immunogenicity of ascending dosages of the vaccine will be assessed. Fifteen subjects will receive vaccine at each of the following dosage levels: 10^8 viral particles (vp)/milliliters (ml), 10^9 vp/ml, 10^10 vp/ml and 10^11 vp/ml with 3 subjects receiving control at each of these dosage levels. Dosage escalation will proceed only after review of the safety data by the Safety Monitoring Committee of the prior dosage level. The primary objective is to assess the safety and reactogenicity of ascending dosages of Adenovirus Type 35 based circumsporozoite malaria vaccine among healthy subjects given in 3 intramuscular doses at 0, 1 and 6 months. The secondary objective is to evaluate the immunogenicity of the Adenovirus Type 35 based circumsporozoite malaria vaccine through performance of Humoral Immune Assays [ELISA (enzyme-linked immunosorbent assay)] for antibodies to circumsporozoite antigen and Adenovirus Neutralization Assay for neutralizing antibodies to Adenovirus type 35) and Cellular Immune Assays [enzyme-linked immunosorbent spot (ELISPOT) and Flow Cytometry] for circumsporozoite (CS)-specific cluster of differentiation (CD)4+ and CD8+ T cell responses.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent before any protocol procedures are performed.
* Males and non-pregnant females between the ages of 18 and 45 years, inclusive.
* Females and males must agree to practice adequate contraception until at least 28 days following their last immunization dose (including abstinence; hormonal contraception; condoms with spermicidal agents; post-menopausal; or surgical sterilization/vasectomy).
* Participants must agree to avoid high risk sexual behavior for exposure to human immunodeficiency virus (HIV).
* In good health as determined by screening medical history, physical examination (PE), and laboratory assessments.
* Willingness to comply with protocol requirements.
* Willingness to be contacted annually for five years for assessment of serious adverse events.
* Must have access to a cell phone.

Exclusion Criteria:

* Current or recent (within the last four weeks) treatment with parenteral, inhaled, or oral corticosteroids (intranasal steroids are acceptable), or other immunosuppressive agents, or chemotherapy.
* History of splenectomy.
* Abnormal screening laboratory values. Any abnormal screening value for any screening test will exclude the subject from the study. Abnormal screening labs will not be repeated with the exception of high glucose levels will be repeated at a fasting state.
* Detectible neutralizing antibody titer against adenovirus serotype 35.
* History of intravenous (IV) drug abuse.
* History of, or current medical, occupational, social or family problems as a result of alcohol or illicit drug use.
* History of moderate to severe mental illness, as defined by symptoms interfering with social or occupational function or suicidal thoughts/attempts.
* History of receiving blood or blood products (such as blood transfusion, platelet transfusion, immunoglobulins, hyperimmune serum) in the previous 6 months.
* Vaccination with a live vaccine within the past 30 days or with a nonreplicating, inactivated, or subunit vaccine within the last 14 days.
* Known hypersensitivity to components of the vaccine.
* History of acute or chronic medical conditions including, but not limited to, disorders of the liver, kidney, lung, heart, or nervous system, or other metabolic or autoimmune/inflammatory conditions.
* History of coagulation defect or bleeding from (bruising at) multiple sites that cannot be linked to trauma or surgery.
* History of anaphylaxis or severe hypersensitivity reaction.
* Severe asthma, as defined by an emergency room visit or hospitalization within the last 12 months.
* Pregnant or breastfeeding women.
* Acute illness, including temperature greater than 100 degrees Fahrenheit within one week prior to vaccination.
* Positive serology for human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B surface antigen (HBsAg).
* Concurrent participation in other investigational protocols or receipt of an investigational product within the previous 30 days or planned receipt of an investigational product within 28 days following the last immunization dose.
* Identification of any condition that, in the opinion of the investigator, would affect the ability of the subject to understand or comply with the study protocol or would jeopardize the safety or rights of a subject participating in the study.
* History of malignancy, including hematologic and skin cancers (except for a localized basal cell carcinoma), or known immunodeficiency syndrome.
* History of malaria infection or previous receipt of a malaria vaccine.
* History of travel to malaria-endemic area or receipt of antimalarial prophylaxis in the past 12 months.
* Planned travel to a malaria-endemic area prior to Visit 16 (Day 208).
* Pre-medication with analgesic or antipyretic agents in the 6 hours prior to vaccination, or planned medication with analgesic or antipyretic in the 24 hours following vaccination. This criterion should not preclude subjects receiving such medication if the need arises.
* Receipt of a recombinant adenovirus vector vaccine in a prior study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2007-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of local, systemic, and safety laboratory adverse events. | Enrollment through to Day 208

SECONDARY OUTCOMES:
T cell responses against the malaria circumsporozoite antigen by enzyme-linked immunosorbent spot (ELISPOT) and flow cytometry. | Days 28, 56, 120, 180, 208.
Antibody titers against the malaria circumsporozoite antigen via enzyme-linked immunosorbent assay (ELISA). | Days 28, 56, 120, 180, 208.
Neutralizing antibody titers against Adenovirus type 35 by Adenovirus Neutralization Assay. | Days 28, 56, 120, 180, 208.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Stanford University School of Medicine, Stanford, California
  - Vanderbilt University - Pediatric - Vanderbilt Vaccine Research Center, Nashville, Tennessee